CLINICAL TRIAL: NCT05115123
Title: Duloxetine Efficacy and Tolerability for Pain Management in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Duloxetine for Postoperative Pain of Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Collaborators: National Hepatology & Tropical Medicine Research Institute (Other Government)
Responsible Party: Principal Investigator, Noha Mansour, Lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23-2021
Record Dates: First submitted 2021-11-01; First posted 2021-11-10 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): patients scheduled for elective LC will receive 60 mg duloxetine before surgery
  Interventions: Drug: Duloxetine
- Control (Placebo Comparator): patients scheduled for elective LC will receive placebo before surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — 60 mg duloxetine
  Arms: Intervention
Drug: Placebo — Placebo
  Arms: Control

SUMMARY:
Recent studies on the impact of perioperative duloxetine for treatment of acute postoperative pain have yielded positive outcomes with respect to reduction opioid consumption. The aim of the present study is to investigate the role of perioperative duloxetine on the management of postoperative pain in patients undergoing LC.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who are scheduled to undergo elective LC

Exclusion Criteria:

1- Patients with acute pancreatitis 2. Patients undergoing chronic pain treatment 3. Patients who received analgesics or sedatives 24 h before scheduled surgery 3. Patients had alcohol or drug addiction 4. Severe hepatic and renal dysfunction 5. Previous allergic response to duloxetine 6. Pregnancy and lactation 7. Patients with communication problems, cognitive dysfunction, or psychological disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change in postoperative pain between the two groups using visual analogue score (VAS) | 24 Hours postoperative
  pain will be assessed using visual analogue score (VAS) 0-100 mm (0 indicated no pain, 100 denoted the most severe pain)

SECONDARY OUTCOMES:
Postoperative nausea and vomiting (PONV) | 24 Hours postoperative
  will be assessed using PONV scale a 4-point scale: none (0): no nausea, vomiting, and retching; mild (1): happened once; moderate (2): happened 2-3 times; and severe (3): continuous or more than three times.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mansour NO, Boraii S, Elnaem MH, Elrggal ME, Omar T, Abdelraouf A, Abdelaziz DH. Evaluation of preoperative duloxetine use for postoperative analgesia following laparoscopic cholecystectomy: A randomized controlled trial. Front Pharmacol. 2022 Sep 29;13:944392. doi: 10.3389/fphar.2022.944392. eCollection 2022. PMID 36249765